CLINICAL TRIAL: NCT07316608
Title: A Phase I, Randomized, Open-label, 3 or 4-period, 7-treatment, Single-dose, Two Cohort, Crossover Study to Assess the Relative Bioavailability of Laroprovstat/Rosuvastatin Fixed Combination Drug Products to the Single Therapy Products in Healthy Adults
Brief Title: A Phase I, Open-label, Crossover Study Comparing the Relative Bioavailability of a Fixed-Dose Combination of Laroprovstat/Rosuvastatin vs Their Single Therapy Products in Healthy Adults
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D7961C00005
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Healthy Participants
Keywords: Hyperlipidemia; Dyslipidemia; Relative Bioavailability; Pharmacokinetics; Food effect; Fixed combination drug products; Single therapy products; Oral formulations
MeSH Terms: conditions — Hyperlipidemias; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1 Treatment A (Experimental): Participants will receive a single oral Fixed Combination Drug Product (FCDP) test formulation 1 of Dose X laroprovstat/Dose 1 rosuvastatin following an overnight fast.
  Interventions: Drug: Laroprovstat Dose X/Rosuvastatin Dose 1 FCDP test formulation 1
- Cohort 1 Treatment B (Experimental): Participants will receive a single oral FCDP test formulation 2 of Dose X laroprovstat/Dose 1 rosuvastatin following an overnight fast.
  Interventions: Drug: Laroprovstat Dose X/Rosuvastatin Dose 1 FCDP test formulation 2
- Cohort 1 Treatment C (Experimental): Participants will receive a single oral Dose X laroprovstat and a single oral Dose 1 rosuvastatin as Single Therapy Product (STP) reference formulations following an overnight fast.
  Interventions: Drug: Laroprovstat Dose X STP; Drug: Rosuvastatin Dose 1 STP
- Cohort 2 Treatment D (Experimental): Participants will receive a single oral FCDP test formulation 1 of Dose X laroprovstat/Dose 2 rosuvastatin following an overnight fast.
  Interventions: Drug: Laroprovstat Dose X/Rosuvastatin Dose 2 FCDP test formulation 1
- Cohort 2 Treatment E (Experimental): Participants will receive a single oral FCDP test formulation 2 of Dose X laroprovstat/Dose 2 rosuvastatin following an overnight fast.
  Interventions: Drug: Laroprovstat Dose X/Rosuvastatin Dose 2 FCDP test formulation 2
- Cohort 2 Treatment F (Experimental): Participants will receive a single oral Dose X laroprovstat and a single oral Dose 2 rosuvastatin as STP reference formulations following an overnight fast.
  Interventions: Drug: Laroprovstat Dose X STP; Drug: Rosuvastatin Dose 2 STP
- Cohort 2 Treatment G (Experimental): Participants will receive a single oral FCDP test formulation 1 of Dose X laroprovstat/Dose 2 rosuvastatin in a fed state.
  Interventions: Drug: Laroprovstat Dose X/Rosuvastatin Dose 2 FCDP test formulation 1

INTERVENTIONS:
Drug: Laroprovstat Dose X/Rosuvastatin Dose 1 FCDP test formulation 1 — Laroprovstat Dose X/Rosuvastatin Dose 1 FCDP test formulation 1 will be administered as an oral tablet in the morning on Day 1 of a given treatment period.
  Arms: Cohort 1 Treatment A
Drug: Laroprovstat Dose X/Rosuvastatin Dose 2 FCDP test formulation 1 — Laroprovstat Dose X/Rosuvastatin Dose 2 FCDP test formulation 1 will be administered as an oral tablet in the morning on Day 1 of a given treatment period.
  Arms: Cohort 2 Treatment D; Cohort 2 Treatment G
Drug: Laroprovstat Dose X/Rosuvastatin Dose 1 FCDP test formulation 2 — Laroprovstat Dose X/Rosuvastatin Dose 1 FCDP test formulation 2 will be administered as an oral tablet in the morning on Day 1 of a given treatment period.
  Arms: Cohort 1 Treatment B
Drug: Laroprovstat Dose X/Rosuvastatin Dose 2 FCDP test formulation 2 — Laroprovstat Dose X/Rosuvastatin Dose 2 FCDP test formulation 2 will be administered as an oral tablet in the morning on Day 1 of a given treatment period.
  Arms: Cohort 2 Treatment E
Drug: Laroprovstat Dose X STP — Laroprovstat Dose X STP will be administered as an oral tablet in the morning on Day 1 of a given treatment period.
  Arms: Cohort 1 Treatment C; Cohort 2 Treatment F
Drug: Rosuvastatin Dose 1 STP — Rosuvastatin Dose 1 STP will be administered as an oral tablet in the morning on Day 1 of a given treatment period.
  Arms: Cohort 1 Treatment C
Drug: Rosuvastatin Dose 2 STP — Rosuvastatin Dose 2 STP will be administered as an oral tablet in the morning on Day 1 of a given treatment period.
  Arms: Cohort 2 Treatment F

SUMMARY:
The purpose of this study is to assess how well laroprovstat and rosuvastatin combined in a single tablet to be taken by mouth works compared with laroprovstat and rosuvastatin individual tablets taken by mouth (relative bioavailability) in healthy adults.

DETAILED DESCRIPTION:
This is a randomized, open-label, 3 or 4-period, single-dose, two-cohort, multi-center, crossover study. The study will comprise of a screening period (21 Days), 3 or 4 treatment periods (depending on cohort assignment) and washout period (14 Days, starting after dosing on Study Day 1 of a given treatment period). Each treatment period consists of dosing on Day 1; any subsequent treatment period will not start sooner than 14 days following dosing in the previous treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study-specific procedures.
* Healthy male and female participants aged 18 to 55 years (inclusive) with suitable veins for cannulation or repeated venipuncture.
* All females must have a negative pregnancy test at the Screening Visit and on admission to the Clinical Unit.
* Females of childbearing potential must not be lactating and if heterosexually active must agree to use an approved method of highly effective contraception, in addition to a barrier method, to avoid pregnancy from the time of first administration of study intervention until 10 days after discharge from the study site.
* Females of non-childbearing potential must be confirmed at the Screening Visit by checking if they are postmenopausal [amenorrhea for at least 12 months following cessation of all exogenous hormonal treatments and follicle stimulating hormone (FSH) levels in the postmenopausal range] or by documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy but not tubal ligation or tubal occlusion.
* Have a body mass index between 18 and 30 kg/m2 inclusive and weigh at least 50 kg.

Exclusion Criteria:

* History of any clinically important disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any prior gastrointestinal surgery which may affect absorption, example (eg), gastric bypass or resection.
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of study intervention.
* Asian origin.
* Any laboratory values with the following deviations at the Screening Visit or on admission to the study site. Abnormal values may be repeated once at the discretion of the investigator:

  * ALT > upper limit of normal (ULN).
  * AST > ULN.
  * TBL > ULN.
  * Estimated glomerular filtration rate < 90 mL/min/1.73 m2 calculated using the Chronic Kidney Disease Epidemiology Collaboration equation.
  * Hemoglobin < lower limit normal (LLN).
  * Creatine kinase > 5 × ULN.
* Inadequately treated hypothyroidism defined as TSH > 1.5 × ULN at screening or participants whose thyroid replacement therapy was initiated or modified within the last 3 months prior to screening.
* Any clinically important abnormalities in clinical chemistry, hematology, or urinalysis results other than those listed above, at screening and/or admission to the study site, as judged by the investigator. Abnormal values may be repeated once at the discretion of the investigator.
* Any positive result on screening for serum Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (HBcAb), Hepatitis C virus (HCV), or Human immunodeficiency virus (HIV).
* Abnormal vital signs, after 10 minutes supine rest, at the Screening Visit and/or admission to the study site, defined as any of the following. Abnormal values may be repeated once (one triplicate measurement) at the discretion of the investigator:

  * Systolic Blood pressure (BP) < 90 mmHg or ≥ 140 mmHg.
  * Diastolic BP < 50 mmHg or ≥ 90 mmHg.
  * Pulse rate < 45 or > 90 beats per minute (bpm).
* Any clinically significant abnormalities on 12-lead electrocardiogram (ECG) at screening and/or admission to the study site, as judged by the investigator. Abnormal values may be repeated once at the discretion of the investigator.
* Current smokers or those who have smoked or used nicotine products (including e cigarettes) within the previous 3 months prior to screening.
* Known or suspected history of alcohol or drug abuse or excessive intake of alcohol as judged by the investigator in the last one year.
* Positive screen for drugs of abuse, alcohol, or cotinine at screening or on each admission to the study site.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to laroprovastat or rosuvastatin.
* Excessive intake of caffeine-containing drinks or food (eg, coffee, tea, chocolate) defined as the regular consumption of more than 500 mg of caffeine per day (eg, > 5 cups of coffee [one cup ~100 mg caffeine]; one cup of tea ~30 mg caffeine) or would likely be unable to refrain from the use of caffeine-containing beverages during confinement at the study site.
* Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks prior to the first administration of study intervention.
* Use of any prescribed or nonprescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, intake of > 3 × daily recommended levels of vitamins and minerals during the 2 weeks prior to the first administration of study intervention or longer if the medication has a long half-life. Hormonal contraceptives (for females of childbearing potential) are allowed.
* Treatment with any lipid lowering therapy or laroprovastat within the 3 months prior to the Screening Visit.
* Treatment with drugs for reduction or inhibition of Proprotein convertase subtilisin/kexin type 9 (PCSK9) within the last 12 months prior to the Screening Visit (approved or investigational and apart from laroprovstat).
* Current or previous administration of inclisiran.
* Plasma donation within one month of the Screening Visit or any blood donation/blood loss > 500 mL during the 3 months prior to the Screening Visit.
* Has received any Investigational Medicinal Product (IMP-defined as a compound which has not been approved for marketing) within 30 days or 5 half-lives (whichever is longest) of the first administration of study intervention in this study.
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
* Judgment by the investigator that the participant should not participate in the study if they have any ongoing or recent (ie, during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
* Participants who have medical dietary restrictions or are unable/unwilling to comply with the meals provided in the unit during the stay at the study site.
* Participants who cannot communicate reliably with the investigator.
* Vulnerable participants, eg, kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-03-16 (Estimated); Primary Completion 2026-05-25 (Estimated); Study Completion 2026-05-25 (Estimated)

PRIMARY OUTCOMES:
Area under concentration time curve from time 0 to infinity (AUCinf) | At predefined intervals from Day 1 to Day 11
  To evaluate the relative bioavailability between the FCDP test formulation 1 and the STPs of laroprovstat and rosuvastatin across the planned rosuvastatin dose range, Dose 1 (Cohort 1) to Dose 2 (Cohort 2)
Area under concentration curve from time 0 to the last quantifiable concentration (AUClast) | At predefined intervals from Day 1 to Day 11
  To evaluate the relative bioavailability between the FCDP test formulation 1 and the STPs of laroprovstat and rosuvastatin across the planned rosuvastatin dose range, Dose 1 (Cohort 1) to Dose 2 (Cohort 2).
Maximum observed drug concentration (Cmax) | At predefined intervals from Day 1 to Day 11
  To evaluate the relative bioavailability between the FCDP test formulation 1 and the STPs of laroprovstat and rosuvastatin across the planned rosuvastatin dose range, Dose 1 (Cohort 1) to Dose 2 (Cohort 2)

SECONDARY OUTCOMES:
Terminal rate constant (λz) | At predefined intervals from Day 1 to Day 11
  To examine the PK profiles of laroprovstat and rosuvastatin when administered as FCDP test formulation 1 or STPs.
Time to reach maximum observed concentration (tmax) | At predefined intervals from Day 1 to Day 11
  To examine the PK profiles of laroprovstat and rosuvastatin when administered as FCDP test formulation 1 or STPs.
Terminal elimination half life (t1/2λz) | At predefined intervals from Day 1 to Day 11
  To examine the PK profiles of laroprovstat and rosuvastatin when administered as FCDP test formulation 1 or STPs.
Apparent total body clearance (CL/F) | At predefined intervals from Day 1 to Day 11
  To examine the PK profiles of laroprovstat and rosuvastatin when administered as FCDP test formulation 1 or STPs.
Apparent volume of distribution based on the terminal phase (V/F) | At predefined intervals from Day 1 to Day 11
  To examine the PK profiles of laroprovstat and rosuvastatin when administered as FCDP test formulation 1 or STPs.
AUCinf | At predefined intervals from Day 1 to Day 11
  To examine the effect on the PK profiles of laroprovstat and rosuvastatin when administered as an FCDP test formulation 1 with high fat meal compared to when administered as an FCDP test formulation 1 in the fasted state.
AUClast | At predefined intervals from Day 1 to Day 11.
  To examine the effect on the PK profiles of laroprovstat and rosuvastatin when administered as an FCDP test formulation 1 with high fat meal compared to when administered as an FCDP test formulation 1 in the fasted state.
Cmax | At predefined intervals form Day 1 to Day 11
  To examine the effect on the PK profiles of laroprovstat and rosuvastatin when administered as an FCDP test formulation 1 with high fat meal compared to when administered as an FCDP test formulation 1 in the fasted state.
tmax | At predefined intervals from Day 1 to Day 11
  To examine the effect on the PK profiles of laroprovstat and rosuvastatin when administered as an FCDP test formulation 1 with high fat meal compared to when administered as an FCDP test formulation 1 in the fasted state.
λz | At predefined intervals form Day 1 to Day 11
  To examine the effect on the PK profiles of laroprovstat and rosuvastatin when administered as an FCDP test formulation 1 with high fat meal compared to when administered as an FCDP test formulation 1 in the fasted state.
t1/2λz | At predefined intervals from Day 1 to Day 11.
  To examine the effect on the PK profiles of laroprovstat and rosuvastatin when administered as an FCDP test formulation 1 with high fat meal compared to when administered as an FCDP test formulation 1 in the fasted state.
CL/F | At predefined intervals form Day 1 to Day 11
  To examine the effect on the PK profiles of laroprovstat and rosuvastatin when administered as an FCDP test formulation 1 with high fat meal compared to when administered as an FCDP test formulation 1 in the fasted state.
V/F | At predefined intervals from Day 1 to Day 11
  To examine the effect on the PK profiles of laroprovstat and rosuvastatin when administered as an FCDP test formulation 1 with high fat meal compared to when administered as an FCDP test formulation 1 in the fasted state.

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- See also: TY card — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7961C00005&attachmentIdentifier=84bce86f-7c45-4029-a976-98797f0aa9da&fileName=AZ_D7961C00005_TY_v1.0_A4_2025_12_15.pdf&versionIdentifier=